CLINICAL TRIAL: NCT01862003
Title: AZD8931, an Inhibitor of EGFR, ERBB2 and ERBB3 Signalling, in Combination With FOLFIRI: a Phase I/II Study to Determine the Importance of Schedule and Activity in Colorectal Cancer
Brief Title: Phase I/II Trial of Antagonism of HER in GI Cancer
Acronym: PANTHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0136
Record Dates: First submitted 2013-05-07; First posted 2013-05-24 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Colorectal Cancer; Recurrent Colorectal Cancer
Keywords: Colorectal cancer; Metastatic Colorectal cancer; Recurrent Colorectal cancer; FOLFIRI; AZD8931; Chemotherapy; EGFR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — AZD 8931; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): AZD8931 160 mg bd, on days 1-4, + FOLFIRI in a 2 weekly schedule
  Interventions: Drug: AZD8931; Drug: Irinotecan; Drug: Folinic Acid; Drug: Fluorouracil

INTERVENTIONS:
Drug: AZD8931 — 160 mg AZD8931 tablets, twice daily on days 1 - 4 of each 2-weekly cycle
Drug: Irinotecan — 180 mg/m2 (IV infusion) of Irinotecan on day 1 of each 2-weekly cycle - can be given simultaneously with Folinic acid.
Drug: Folinic Acid — 350 mg (IV infusion) of Folinic acid on day 1 of each 2-weekly cycle - can be given simultaneously with Irinotecan.
Drug: Fluorouracil — 400 mg/m2 (IV bolus) of Fluorouracil on day 1 of each 2-weekly cycle, to be given after completion of Irinotecan and Folinic acid.
Drug: Fluorouracil — 2400 mg/m2 (IV) continuous infusion of Fluorouracil given over 46 hours - infusion to start after 5FU bolus.

SUMMARY:
Recruitment to phase I of the PANTHER trial is complete.

Phase II, is to evaluate the best overall response rate for AZD8931 + FOLFIRI treatment.

DETAILED DESCRIPTION:
PANTHER is a registered phase I/phase II trial in patients with recurrent or metastatic colorectal cancer.

The phase II part of the study will be a single arm trial. Patients will receive AZD8931 (an EGFR/ERBB inhibitor) in combination with FOLinic acid, Fluorouracil and IRInotecan (FOLFIRI), Treatment will be given in two-weekly cycles. Phase II's primary objective is to evaluate the Best overall response

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological/cytological diagnosis of non-resectable, recurrent or metastatic colorectal cancer
2. Tumour with wild-type RAS
3. Measurable disease evaluated by RECIST criteria v1.1
4. WHO performance status 0 or 1
5. Age ≥ 16
6. Estimated life expectancy > 3 months
7. Adequate haematological function:

   * Haemoglobin ≥100 g/L
   * Absolute neutrophil count ≥1.5 x 10^9/L
   * Platelet count ≥100 x 10^9/L
8. Adequate liver function:

   * Total bilirubin ≤1.5 x upper limit of normal (ULN) (except for patients with known documented cases of Gilbert's syndrome)
   * ALT, AST & ALP ≤2.5 x ULN in the absence of noted liver metastases
   * ALT, AST & ALP ≤5 x ULN in the presence of liver metastases
9. Adequate renal function:

   * Serum creatinine ≤1.5 x ULN
   * Calculated creatinine clearance ≥30 mL/min
10. Adequate biliary drainage (patients with stents are eligible)
11. Adequate venous access for collection of exploratory biological samples
12. Women of child-bearing potential must have a negative pregnancy test prior to study entry. Female patients and male patients with partners of child-bearing potential must agree to use an adequate contraception method, which must be continued for 6 months after completion of chemotherapy
13. Must be able to swallow AZD8931 tablets
14. Capable of giving written informed consent
15. The following prior therapy is allowed:

    * Surgery - patients may have undergone a non-curative operation or palliative bypass surgery only. Patients who have previously undergone curative surgery must have evidence of non-resectable disease relapse
    * Radiotherapy - for localised disease
    * Prior adjuvant chemotherapy - provided this was completed at least 6 months before trial entry

Exclusion Criteria:

1. Patients undergoing treatment with curative intent
2. Any prior treatment with agents targeting the ERBB pathway
3. Treatment with experimental drugs within 30 days or 5 half-lives of first dose of AZD8931
4. Previous palliative chemotherapy
5. Prior treatment with anthracyclines or mitoxantrone
6. Current disease or condition known to interfere with absorption, distribution, metabolism or excretion of drugs (including refractory nausea and vomiting, chronic gastrointestinal disease (e.g. inflammatory bowel disease), or significant bowel resection)
7. History of prior malignancy that will interfere with the response evaluation (exceptions listed in protocol)
8. Evidence of severe/uncontrolled systemic diseases or laboratory finding that makes it undesirable for the patient to participate in the trial
9. Evidence of active uncontrolled infection
10. Patients with clinically significant ascites and/or effusions
11. Regular use of anti-diarrhoeal
12. Pregnant or lactating women
13. Cardiac conditions (as detailed in the trial protocol)
14. Any psychiatric or other disorder (e.g. brain metastases) likely to impact the ability to give informed consent
15. Eye conditions (as detailed in the trial protocol)
16. Patients with chronic skin conditions e.g. acne rosacea, psoriasis, severe atopic eczema
17. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
18. History or repeated unexplained episodes of syncope/dizziness
19. Known hypersensitivity to AZD8931, its excipients, or drugs in its class
20. The use of drugs/substances known to inhibit or induce CYP3A4 or CYP2D6, or those known to prolong QT interval, which cannot be discontinued for the duration of trial treatment
21. Patients with hereditary fructose intolerance

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Best overall response | From registration to date of documented best response, assessed up to 36 months
  Best overall response will be assessed according to RECIST v1.1.

SECONDARY OUTCOMES:
To evaluate the efficacy of AZD8931 plus FOLFIRI | Baseline to 12 weeks post treatment start
  Percentage change in tumour size will be considered the best response only if a second assessment has been carried out which confirms SD at least four weeks after trial entry. Assessment will be determined using CT scans performed at baseline, 12 weeks after start of chemotherapy, then every 3 months until disease progression up to 3 years from registration/ randomisation
Progression Free Survival | From date of randomisation to date of documented disease progression or death from any cause, whichever comes first, assessed up to 3 years from date of registration/ randomisation
  Progression-free survival time will be calculated from the date of trial entry to the date of documented progression, or death from any cause. In cases where progression is suspected and subsequently confirmed by scans, the date of documented suspected progression will be used.
Overall Survival | From date of registration/ randomisation until date of death or date of last follow-up assessment (up to 3 years from date of registration/ randomisation)
  Overall survival time will be calculated from the date of trial entry to the date of death from any cause or end of trial follow-up.
Occurrence and Severity of Adverse Events | From date of registration/ randomisation until 30 days after completion of trial treatment (AZD8931 and FOLFIRI)
  Will include all grade 1-5 adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hochhauser, BA, MBBS, MRCP, D.PHIL, FRCP, Principal Investigator — University College London (UCL) Cancer Institute
Locations (4):
- United Kingdom (4):
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University College London Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Propper DJ, Gao F, Saunders MP, Sarker D, Hartley JA, Spanswick VJ, Lowe HL, Hackett LD, Ng TT, Barber PR, Weitsman GE, Pearce S, White L, Lopes A, Forsyth S, Hochhauser D. PANTHER: AZD8931, inhibitor of EGFR, ERBB2 and ERBB3 signalling, combined with FOLFIRI: a Phase I/II study to determine the importance of schedule and activity in colorectal cancer. Br J Cancer. 2023 Jan;128(2):245-254. doi: 10.1038/s41416-022-02015-x. Epub 2022 Nov 9. PMID 36352028